CLINICAL TRIAL: NCT02403401
Title: Multi-center, Open-label, Single-arm Study to Assess the Safety and Contraceptive Efficacy of a Levonorgestrel-containing Intravaginal Ring During a Treatment Period of One Year in Healthy Women 18 to 35 Years of Age
Brief Title: Safety and Contraceptive Efficacy of an Intravaginal Ring With LNG (Levonorgestrel) Over One Year in Healthy Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16803
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Contraception
Keywords: Pregnancy prevention
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levonorgestrel (BAY98-7196) (Experimental): Vaginal ring containing 170 mg levonorgestrel
  Interventions: Drug: Levonorgestrel (BAY98-7196)

INTERVENTIONS:
Drug: Levonorgestrel (BAY98-7196) — Levonorgestrel 40 µg/d intravaginal ring (treatment for 365 days, 28 days wearing period for each ring)

SUMMARY:
Purpose of the study is to investigate safety and contraceptive efficacy of an LNG-containing intravaginal ring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subject requesting contraception and willing to use the IVR
* Normal or clinically insignificant cervical smear not requiring further follow up (a cervical smear has to be taken at screening visit or a normal result has to be documented within the previous 6 months)
* History of regular cyclic menstrual periods
* Subject is willing and able to attend the scheduled study visits and comply with study procedures

Exclusion Criteria:

* Pregnancy or lactation (less than three months since delivery, abortion, or lactation before start of treatment)
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Any disease or condition that may worsen under hormonal treatment according to the assessment and opinion of the investigator
* Undiagnosed abnormal genital bleeding
* Wish for pregnancy during the study
* Major surgery scheduled during the study period

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1471 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate (Pearl Index) | Up to 12 months
  Pearl Index = Number of pregnancies per 100 woman-years of exposure

SECONDARY OUTCOMES:
Cumulative failure rate | Up to 12 months
  Probability of getting pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (86):
- United States (70):
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Mesa, California
  - Sacramento, California
  - San Diego, California
  - Denver, Colorado
  - New London, Connecticut
  - Clearwater, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Lake Worth, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - North Miami, Florida
  - Oviedo, Florida
  - St. Petersburg, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Idaho Falls, Idaho
  - Champaign, Illinois
  - Chicago, Illinois
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Johnson City, New York
  - Port Jefferson, New York
  - Rochester, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Myrtle Beach, South Carolina
  - Summerville, South Carolina
  - Jackson, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Draper, Utah
  - Pleasant Grove, Utah
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Japan (16):
  - Funabashi, Chiba
  - Yotsukaidō, Chiba
  - Aki-gun, Hiroshima
  - Sapporo, Hokkaido
  - Kurashiki, Okayama-ken
  - Chuo-ku, Tokyo
  - Hachiōji, Tokyo
  - Nakano-ku, Tokyo
  - Nishitōkyō, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinjuku, Tokyo
  - Toshima-ku, Tokyo
  - Fukui
  - Fukuoka
  - Osaka

REFERENCES:
- [Derived] Nave R, Hochel J, Mellinger U, Kohnke A, Elliesen J, Schmitz H. Pearl Index study with levonorgestrel-releasing intravaginal rings: using pharmacokinetic results to investigate treatment compliance as a potential contributor for contraceptive failure. Hum Reprod. 2020 Nov 1;35(11):2515-2523. doi: 10.1093/humrep/deaa195. PMID 32914172